CLINICAL TRIAL: NCT01993979
Title: A Phase III Randomised Trial of Peri-Operative Chemotherapy Versus sUrveillance in Upper Tract Urothelial Cancer
Brief Title: A Phase III Randomised Trial of Peri-Operative Chemotherapy Versus sUrveillance in Upper Tract Urothelial Cancer (POUT)
Acronym: POUT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICR-CTSU/2011/10031; 2011-002577-33 (EudraCT Number); ISRCTN98387754 (Registry Identifier: ISRCTN); CRUK/11/027 (Other Grant/Funding Number: Cancer Research UK (CR UK)); 11/NW/0782 (Other: Main REC)
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Transitional Cell Carcinoma of Ureter
Keywords: Adjuvant chemotherapy; Surveillance; Nephro-ureterectomy
MeSH Terms: interventions — Drug Therapy; Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surveillance (Other): Patients allocated to surveillance will be seen at 4, 7, 10 and 13 weeks post randomisation - equivalent to the end of cycle in patients receiving chemotherapy - in order to collect details of early treatment failure in this group and comparative data relating to toxicity and quality of life. Patients on surveillance will then be followed up for signs of recurrence at the same intervals as those who received chemotherapy
  Interventions: Other: Surveillance
- Chemotherapy (Experimental): Patients allocated adjuvant chemotherapy will receive 4 x 21 day cycles of gemcitabine-cisplatin. Patients who have a sub-optimal renal function (GFR 30-49ml/min) will receive carboplatin instead of cisplatin.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy
  Other Names: Gemcitabine; Cisplatin; Carboplatin
  Arms: Chemotherapy
Other: Surveillance — Patients will be closely monitored for early signs of recurrence, for which they will receive treatment as decided in discussion between the clinician and patient. This may include chemotherapy.
  Arms: Surveillance

SUMMARY:
POUT is a multi-centred randomised controlled phase III trial. 345 patients who have undergone nephro-ureterectomy, are surgically staged pT2-pT4, N0-3 or are pT1 and node positive, and who are fit for adjuvant chemotherapy, will be randomised to four cycles of adjuvant platinum based chemotherapy (experimental group) or surveillance (control group). Participants will be followed up according to routine practice.

Primary endpoint: Disease-free survival (DFS)

Secondary endpoints:

* Overall Survival
* Metastasis free survival
* Incidence of bladder second primary tumours
* Incidence of contralateral primary tumours
* Acute and late toxicity
* Treatment compliance
* Quality of life

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* ≥18 years of age
* Post radical nephro-ureterectomy for upper tract tumour with predominant TCC component - squamoid differentiation or mixed TCC/SCC is permitted.
* Histologically confirmed TCC staged pT2-pT4 pN0-3 M0 or pTany N1-3 M0 (providing all grossly abnormal nodes are resected). Patients with microscopically positive margins on pathology may be entered (providing all grossly abnormal disease was resected).
* Satisfactory haematological profile (ANC> 1.5 x 109/L, platelet count ≥ 100 x 109/L) and liver function tests (bilirubin < 1.5 x ULN, AST and Alkaline phosphatase < 2.5 x ULN), Glomerular filtration rate ≥30 mls/min.
* Fit and willing to receive adjuvant chemotherapy with first cycle to be commenced within 90 days of radical nephro-ureterectomy if allocated
* WHO performance status 0-1.
* Available for long-term follow-up

Exclusion Criteria:

* Evidence of distant metastases
* Pure adenocarcinoma, squamous cell carcinoma or small cell or other variant histology
* Un-resected macroscopic nodal disease
* Concurrent muscle invasive bladder cancer (patients with concurrent Non-muscle invasive bladder cancer (NMIBC) will be eligible)
* GFR <30 ml/minute. NB Gemcitabine-carboplatin can only be given for patients with suboptimal renal function for cisplatin i.e. for GFR 30-49ml/min. Patients with poor performance status or co-morbidities that would make them unfit for chemotherapy are ineligible for the trial
* Significant co-morbid conditions that would interfere with administration of protocol treatment
* Pregnancy; lactating women or women of childbearing potential unwilling or unable to use adequate non-hormonal contraception (male patients should also use contraception if sexually active);
* Previous malignancy in the last 5 years except for previous NMIBC, adequately controlled non melanoma skin tumours, CIS of cervix or LCIS of breast or localised prostate cancer in patients who have a life expectancy of over 5 years upon trial entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2012-05; Primary Completion 2018-11-07 (Actual); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 3 years
  To determine whether adjuvant combination chemotherapy improves the disease-free survival for patients with resected histologically confirmed muscle invasive (pT2-T4, N0-3) or node positive upper tract TCC.

SECONDARY OUTCOMES:
Overall survival | Patients followed-up for 5 years
  Whether adjuvant platinum-based chemotherapy improves overall survival in this patient group
Metastasis free survival | Patients are followed up for 5 years
  To determine whether adjuvant platinum-based chemotherapy improves metastasis free survival in this patient group.
Incidence of bladder second primary tumours | Patients are followed up for 5 years
  Whether adjuvant platinum-based chemotherapy reduces incidence of second primary urothelial cancers
Incidence of contralateral primary tumours | Patients are followed up for 5 years
  To determine whether adjuvant platinum-based chemotherapy reduces incidence of contralateral primary urothelial cancers.
Acute and late toxicity | Patients are followed up for 5 years
  To assess the toxicity of chemotherapy in this patient group.
Quality of life (QoL) | Patients' QoL will be assessed over 2 years
  To assess the relative quality of life in patients undergoing adjuvant chemotherapy or surveillance in this patient group.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Alison Birtle, Principal Investigator — Lancashire Teaching Hospitals NHS Foundation Trust
Locations (61):
- United Kingdom (61):
  - William Harvey Hospital, Ashford-Kent, England
  - North Devon District Hospital, Barnstaple, England
  - Basildon University Hospital, Basildon, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Royal Free Hospital, Hampstead, London, England
  - Ipswich Hospital NHS Trust, Ipswich, England
  - St. James's University Hospital, Leeds, England
  - Barts and the London School of Medicine, London, England
  - Maidstone Hospital, Maidstone, England
  - Christie Hospital NHS Trust, Manchester, England
  - Queen Elizabeth The Queen Mother Hospital, Margate, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Peterborough Hospitals Trust, Peterborough, England
  - Rosemere Cancer Centre at Royal Preston Hospital, Preston, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Royal Marsden Hosital, Sutton, Surrey, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - New Cross Hospital, Wolverhampton, England
  - Ayr Hospital, Ayr, Scotland
  - Velindre Cancer Center at Velinde Hospital, Cardiff, Wales
  - Singleton Hospital, Swansea, Wales
  - Bristol Haematology and Oncology Centre, Bristol
  - Southmead Hospital, Bristol
  - Royal Marsden Hospital, Chelsea
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Darent Valley Hospital, Dartford
  - Royal Derby Hospital, Derby
  - Royal Bournemouth General Hospital, Dorset
  - Western General Hospital, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Surrey County Hospital, Guildford
  - Calderdale Royal Infirmary, Halifax
  - Huddersfield Royal Infirmary, Huddersfield
  - Caithness General Hospital, Inverness
  - Raigmore Hospital, Inverness
  - Leicester Royal Infirmary, Leicester
  - Lincoln County Hospital, Lincoln
  - Royal Liverpool University Hospital, Liverpool
  - Guy's Hospital, London
  - Charing Cross Hospital, London
  - Northwick Park Hospital, London
  - Manchester Royal Infirmary, Manchester
  - James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle upon Tyne
  - Norfolk and Norwich University Hospital, Norwich
  - Queen Alexandra Hospital,, Portsmouth
  - Glan Clywd Hospital, Rhyl
  - Queen's Hospital,, Romford, Essex
  - Royal Shrewsbury Hospital, Shrewsbury
  - Southampton General Hospital, Southampton
  - Lister Hospital, Stevenage
  - University Hospital of North Tees, Stockton-on-Tees
  - Frimley Park Hospital, Surrey
  - The Royal Marsden Hospital, Sutton
  - Musgrove Park Hospital, Taunton
  - Torbay District General Hospital, Torbay
  - Royal Cornwall Hospital, Treliske
  - Worthing Hospital, Worthing
  - York District Hospital, York

REFERENCES:
- [Result] Birtle A, Johnson M, Chester J, Jones R, Dolling D, Bryan RT, Harris C, Winterbottom A, Blacker A, Catto JWF, Chakraborti P, Donovan JL, Elliott PA, French A, Jagdev S, Jenkins B, Keeley FX Jr, Kockelbergh R, Powles T, Wagstaff J, Wilson C, Todd R, Lewis R, Hall E. Adjuvant chemotherapy in upper tract urothelial carcinoma (the POUT trial): a phase 3, open-label, randomised controlled trial. Lancet. 2020 Apr 18;395(10232):1268-1277. doi: 10.1016/S0140-6736(20)30415-3. Epub 2020 Mar 5. PMID 32145825
- [Derived] Birtle AJ, Jones R, Chester J, Lewis R, Biscombe K, Johnson M, Blacker A, Bryan RT, Catto JWF, Choudhury A, Das P, Jagdev S, Powles T, Wagstaff J, Cheung KC, Cafferty F, Hall E. Improved Disease-Free Survival With Adjuvant Chemotherapy After Nephroureterectomy for Upper Tract Urothelial Cancer: Final Results of the POUT Trial. J Clin Oncol. 2024 May 1;42(13):1466-1471. doi: 10.1200/JCO.23.01659. Epub 2024 Feb 13. PMID 38350047